CLINICAL TRIAL: NCT06942052
Title: Correlation Between Forward Head Posture, Cervical Range of Motion, and Nerve Conduction Values in Carpal Tunnel Cases
Acronym: FHPCTS
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hany Mohamed Ibrahim Elgohary, Professor, Cairo University
Other Study IDs: P.T.REC/012/003566
Record Dates: First submitted 2025-04-15; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: forward head posture; cervical range of motion; nerve conduction velocity
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group consisted of 84 individuals diagnosed with CTS: The study group consisted of 84 individuals diagnosed with CTS, participants exhibiting forward head posture. All participants had a CVA score of less than 49 degrees. NCS were conducted on both groups to gather relevant NCS values, and measurements of cervical ROM were also taken. Additionally, the visual analog scale (VAS) was utilized to evaluate pain levels, and the body mass index (BMI) for each participant was calculated.
- control group included 35 participants: control group included 35 participants exhibiting forward head posture. All participants had a CVA score of less than 49 degrees. NCS were conducted on to gather relevant NCS values, and measurements of cervical ROM were also taken. Additionally, the visual analog scale (VAS) was utilized to evaluate pain levels, and the body mass index (BMI) for each participant was calculated.

SUMMARY:
Before the examination, participants underwent thorough preparation to guarantee the accuracy and reliability of the study's results. Each participant was provided with a comprehensive overview of the assessment procedures, highlighting the importance of the CVA measurements, NCS, cervical ROM evaluations, and the VAS for assessing pain levels. They were advised to come well-rested and to refrain from any activities that could affect their pain levels or overall physical condition on the assessment day. Furthermore, participants were encouraged to wear comfortable attire to facilitate the examination process. Ensuring a supportive environment was essential, allowing participants to feel at ease while discussing their symptoms and experiences, which is vital for collecting accurate data and fostering cooperation throughout the study.

DETAILED DESCRIPTION:
Participants in this study were referred from the neurophysiology unit at Al-Azhar University Hospital in New Damietta, as well as from the outpatient neurology clinic at Cairo University. The research was conducted at the outpatient clinic of the Faculty of Physical Therapy at Horus University in Damietta. Approval for the study was granted by the ethical committee of Cairo University's Faculty of Physical Therapy, with the approval number P.T.REC/012/003566. All participants provided written consent after a comprehensive explanation of the study's objectives, procedures, potential benefits, privacy considerations, and data utilization.

Sample size determination:

In this case-control study, we aimed to investigate the relationship between exposure and the outcome of interest by analyzing a total of 119 participants, divided into two groups: 84 individuals diagnosed with CTS and 35 controls exhibiting forward head posture. The proportions of exposed individuals were calculated, revealing that approximately 28.57% of the control group and 35.29% of the study group were exposed to the risk factor. The odds ratio (OR) was determined to be 1.3625, indicating that the odds of exposure were about 1.36 times higher in the CTS group compared to the controls. The 95% confidence interval for the OR ranged from 0.576 to 3.21, suggesting a positive association between exposure and the outcome, although the interval includes values less than 1, indicating that the association may not be statistically significant. All participants underwent a CVA with scores below 49 degrees, and NCS were performed to gather relevant values. Additionally, cervical ROM measurements were taken, and pain levels were evaluated using the VAS, while BMI was calculated for each participant.

Participants' Selection:

The study included a total of 119 participants, comprising 35 healthy individuals matched for age and sex, as well as 84 patients diagnosed with carpal tunnel syndrome. All participants exhibited FHP. The CTS patients were diagnosed based on medical assessment by neurologist and confirmed by electrophysiological studies (NCS).

Inclusion criteria:

119 Participants aged between 25 and 40 years from both genders were included in this study with the following criteria: (a) Participants reported pain and paresthesia in the median nerve distribution of the hand for a minimum of three months. (b) Symptoms were noted to worsen at night, (c) A positive Phalen sign (d) A positive Tinel sign [8] and (E) abnormal parameter of electrophysiological studies include prolonged distal motor latency exceeded 4.2 ms and prolonged distal sensory latency exceeded 3.6 ms.

Exclusion criteria:

Participants who had any of the following symptoms were excluded: individuals with current ulnar or radial nerve neuropathy. Previous injection or release for carpal tunnel. Patients with various upper extremity or cervical diseases, such as cervical radiculopathy. Diabetic patients and pregnant females. Patients who had previously undergone cervical surgery had a history of cervical fractures or trauma or had temporomandibular disorders. Patients on antiepileptic medication for neuropathic pain, those with inflammatory or uncontrolled systemic disorders that cause neuropathy.

Procedures:

Before the examination, participants underwent thorough preparation to guarantee the accuracy and reliability of the study's results. Each participant was provided with a comprehensive overview of the assessment procedures, highlighting the importance of the CVA measurements, NCS, cervical ROM evaluations, and the VAS for assessing pain levels. They were advised to come well-rested and to refrain from any activities that could affect their pain levels or overall physical condition on the assessment day. Furthermore, participants were encouraged to wear comfortable attire to facilitate the examination process. Ensuring a supportive environment was essential, allowing participants to feel at ease while discussing their symptoms and experiences, which is vital for collecting accurate data and fostering cooperation throughout the study.

Demographic data collection:

The demographic data were collected, including age, sex, weight, height, and body mass index BMI. BMI was calculated using the following equation: (Weight (Kg))/(Height (m^2))

Assessment of pain intensity using the VAS:

The participants were directed to draw a mark on a 10 cm line. This line shows a scale from no pain (zero) to the worst pain the patient could experience (ten). The patients' pain intensity was determined by recording measurements from the scale's zero point to their marks. [13] VAS scores of 3.4 or lower were classified as mild pain, scores ranging from 3.5 to 7.4 indicated moderate pain, and scores of 7.5 or higher were categorized as severe pain.

Assessment of CTS using phalen test:

A positive Phalen sign was present, indicating that symptoms intensified when the wrists were flexed for a specific duration (2 MIN) if numbness appear in 10 sec this means sever CTS, if numbness appear after 30 sec to 1min. means moderate, if symptoms appear after 1min. mean mild CTS.

Assessment of CTS using Tinel sign:

A positive Tinel sign was also observed when tapping over the median nerve at the wrist, which elicited tingling or pain in the median nerve distribution of the hand mainly palmar surface of lateral 3.5 fingers.

Assessment of cervical range of motion using CROM device:

The participants were guided to sit up straight in a comfortable position with their heads in a neutral position by looking straight forward. Only the head should be moved during the assessment, from forward to backward (flexion and extension), right/left rotation, and right/left lateral flexion, as far as they could do so without experiencing any pain. Three measurements were taken for each motion, and the mean was calculated for the statistical tests.

Assessment of forward head posture:

The forward head position was evaluated by photographing the participants' cervical region from the side and measuring the CVA. A plastic-colored marker was attached directly over the C7 vertebra's spinous process, and the tragus of the ear was marked. The camera was positioned 1.5 meters away from the participants on a stationary base without rotation or tilt, with the base set at the participants' shoulder height. To standardize the participants' neck posture, a self-balanced position was selected. The participants were told to keep their arms by their sides and to focus their vision on a point on the wall directly ahead of them.

In the current study, the CVA was calculated using the Kinovea software by measuring the angle between a line that runs from the tragus of the ear to C7 and a horizontal line that passes through C7. A smaller CVA suggested a higher FHP. The forward head position was considered if the CVA was less than 49 degrees.

Nerve conduction studies:

A neurophysiologist evaluated the electrophysiological results using the Neuropack Nihon Kohden Electrodiagnostic system at Al-Azhar University in New Damietta's Neurophysiology Department. Using standardized techniques, conduction tests of the median nerve were evaluated in both upper extremities. Nerve conduction values were obtained; CTS was defined as sensory distal latency (SDL) of 3.6 ms or more, sensory nerve conduction velocity (SNCV) is 45 m/sec or less, or motor distal latency (MDL) is 4.2 ms or more, and Motor nerve conduction velocity (MNCV) is 45 m/s or less.

Motor conduction studies:

The active recording electrode was placed directly over the thenar muscle (the belly of the abductor pollicis brevis muscle), the reference electrode was placed on the bony prominence at the base of the thumb. The ground electrode was firmly fixed on the dorsum of the hand, between the active and stimulating electrodes.

Distal stimulation was performed at the wrist between the flexor carpi radialis and palmaris longus tendons. Proximal stimulation was performed proximal and medial to the antecubital space medial to the bicep's tendon. The stimulator was placed immediately lateral to the brachial artery to reduce the chance of accidentally electro-stimulating the ulnar nerve.

Sensory conduction studies (Antidromic):

Ring electrodes were used. The active electrode was attached to the proximal segment of the index finger. The reference electrode was positioned on the distal phalanx 3 to 4 cm away from the active electrode. The ground was placed on the dorsal aspect of the hand between the active and stimulating electrodes. Ring electrodes are designed to provide a stable and consistent contact area for recording sensory nerve action potentials. Unlike surface electrodes, which may have variable contact quality, ring electrodes ensure uniform pressure and positioning, which can enhance the accuracy of the measurements. Stimulation was performed at the wrist in the same way as the motor conduction studies.

ELIGIBILITY:
Inclusion Criteria:

* 25 and 40 years
* both genders
* Participants reported pain and paresthesia in the median nerve distribution of the hand for a minimum of three months.
* Symptoms were noted to worsen at night
* A positive Phalen sign
* A positive Tinel sign
* abnormal parameter of electrophysiological studies include prolonged distal motor latency exceeded 4.2 ms and prolonged distal sensory latency exceeded 3.6 ms.

Exclusion Criteria:

* individuals with current ulnar or radial nerve neuropathy.
* Previous injection or release for carpal tunnel.
* Patients with various upper extremity or cervical diseases, such as cervical radiculopathy.
* Diabetic patients
* pregnant females.
* Patients who had previously undergone cervical surgery had a history of cervical fractures or trauma or had temporomandibular disorders.
* Patients on antiepileptic medication for neuropathic pain
* those with inflammatory or uncontrolled systemic disorders that cause neuropathy.

Ages: 22 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 119 Participants aged between 25 and 40 years from both genders were included in this study with the following criteria: (a) Participants reported pain and paresthesia in the median nerve distribution of the hand for a minimum of three months. (b) Symptoms were noted to worsen at night, (c) A positive Phalen sign (d) A positive Tinel sign [8] and (E) abnormal parameter of electrophysiological studies include prolonged distal motor latency exceeded 4.2 ms and prolonged distal sensory latency exceeded 3.6 ms.
Sampling Method: Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2022-06-12 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
visual analogue scale | at the baseline
  The participants were directed to draw a mark on a 10 cm line. This line shows a scale from no pain (zero) to the worst pain the patient could experience (ten). The patients' pain intensity was determined by recording measurements from the scale's zero point to their marks. VAS scores of 3.4 or lower were classified as mild pain, scores ranging from 3.5 to 7.4 indicated moderate pain, and scores of 7.5 or higher were categorized as severe pain.

SECONDARY OUTCOMES:
phalen test | at the baseline
  A positive Phalen sign was present, indicating that symptoms intensified when the wrists were flexed for a specific duration (2 MIN) if numbness appear in 10 sec this means sever CTS, if numbness appear after 30 sec to 1min. means moderate, if symptoms appear after 1min. mean mild CTS.
Tinel sign | measurements were obtained at the time f the study
  A positive Tinel sign was also observed when tapping over the median nerve at the wrist, which elicited tingling or pain in the median nerve distribution of the hand mainly palmar surface of lateral 3.5 fingers.
forward head posture | at the baseline
  The forward head position was evaluated by photographing the participants' cervical region from the side and measuring the CVA. A plastic-colored marker was attached directly over the C7 vertebra's spinous process, and the tragus of the ear was marked. The camera was positioned 1.5 meters away from the participants on a stationary base without rotation or tilt, with the base set at the participants' shoulder height. To standardize the participants' neck posture, a self-balanced position was selected. The participants were told to keep their arms by their sides and to focus their vision on a point on the wall directly ahead of them.
  In the current study, the CVA was calculated using the Kinovea software by measuring the angle between a line that runs from the tragus of the ear to C7 and a horizontal line that passes through C7. A smaller CVA suggested a higher FHP. The forward head position was considered if the CVA was less than 49 degrees.
Nerve conduction studies | at the baseline
  A neurophysiologist evaluated the electrophysiological results using the Neuropack Nihon Kohden Electrodiagnostic system at Al-Azhar University in New Damietta's Neurophysiology Department. Using standardized techniques, conduction tests of the median nerve were evaluated in both upper extremities. Nerve conduction values were obtained; CTS was defined as sensory distal latency (SDL) of 3.6 ms or more, sensory nerve conduction velocity (SNCV) is 45 m/sec or less, or motor distal latency (MDL) is 4.2 ms or more, and Motor nerve conduction velocity (MNCV) is 45 m/s or less.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
it will be available when needed

REFERENCES:
- [Background] Elfahl AM, Abd El Baky AM, Yousef MT, Elgohary HM. High Versus Low Frequency Transcutaneous Electric Nerve Stimulation On Chronic Venous Lower Limb Ulceration Randomized Controlled Trial. Int J Low Extrem Wounds. 2025 Jun;24(2):376-382. doi: 10.1177/15347346221093860. Epub 2022 Apr 14. PMID 35422171